CLINICAL TRIAL: NCT05289076
Title: Protocol for Evaluation of Oncological Treatment in Patients With CRLM Using Zebra Fish Avatars-may This Model Improve Resection Rates and Survival in Patients With Upfront Non-resectable Metastatic Disease?
Brief Title: Evaluation of Tumour Growth and Oncological Treatment in Patients With CRLM Using Zebra Fish Embryo Model
Acronym: CRLM-Z
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Linkoeping (Other)
Collaborators: Medical Research Council of Southeast Sweden (Other Government); Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Per Sandström, Professor of surgery, University Hospital, Linkoeping
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Academic study
Record Dates: First submitted 2022-03-09; First posted 2022-03-21 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Colorectal Cancer Metastatic; Tumour Metastasis; Chemotherapy Effect; Tumor Growth
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Colorectal liver metastsis, single arm (Experimental): Tumour tissue from patients operated for colorectal liver metastases. A cubic centimeter of tumour tissue will be processed and implanted in zebra fish embryos. Tissue in zebrafish embryos will treated with different combinations of chemotherapy. Chemocombination of best effect will be offered patients in the third phase of the trial
  Interventions: Drug: Chemotherapy drug

INTERVENTIONS:
Drug: Chemotherapy drug — Different combinations of chemotherapies will be tested in combination with monoclonal antibodies in zebrafish embryos against inplanted patients livermetastatic tissues.

SUMMARY:
In order to improve and individualize cancer treatment, personalized treatment needs to be developed much further. Liver metastasizing colorectal cancer is treated with a combination of oncological and surgical interventions. The selection of chemotherapy is today mainly done according to best guess. Today only a small fraction of oncological treatment may be known to be effective in a person before treatment start, most often it is trial and error. A fast reliable system for looking at response to different treatments in each unique patient is much needed and would, if successful, completely change the way we give oncological treatment today. Patient's tumor tissue will be evaluated with use of zebrafish embryo avatars to evaluate tumour growth and response to different combinations of chemotherapy. If successful interventional studies are planned.

DETAILED DESCRIPTION:
The possibilities to predict oncological tumor response for individual patients with GI malignancies in order to tailor a personalized oncological treatment, are currently limited. This means that most of the information used to decide upon oncological treatment pertains to a group of patients rather than individuals. Similarly, most of the chemotherapy regimens used is not individually tailored although it has been shown to be beneficial for certain cohorts of patients. In colorectal cancer, KRAS (Kirsten rat sarcoma) and BRAF mutation status predict the response to drugs targeting various steps in the EGFR/KRAS/BRAF signaling pathway, whereas MSI/MMR status may predict the outcome of immune checkpoint inhibitors [1]. As chemotherapy, as well as other cancer treatments, may have severe side effects the treatment may not only be ineffective but may also cause severe adverse events even shortening the patient's life and inhibit the chance of curative tumor resection. For this reason, pre-treatment response evaluation in an avatar model of zebrafish, would be most valuable.

From a clinical point of view the easiest situation is in the adjuvant setting. At this point the whole tumor is available for analysis and larger pieces of tissues may be used in the avatar model. 5-fluorouracil or capecitabine (a 5-FU prodrug) either alone or in combination with oxaliplatin is the current standard adjuvant treatment in stage III colon cancer and stage II colon cancers with 2+ risk factors. Other types of combination regimens including e.g. irinotecan have so far failed to show benefit in the adjuvant situation.

In the neoadjuvant setting, i.e. preoperative treatment to patients with resectable CRLM, combinations of 5-FU (or capecitabine) and either oxaliplatin or irinotecan may improve the outcome of surgery and long term prognosis. It is currently not known which regimen is most efficient for the individual patient.

In the most severe scenario, where the patient presents with unresectable CRLM, either palliative chemotherapy or downsizing/conversion chemotherapy is indicated. For the latter group of patients, it is of uttermost importance to provide as potent treatment as possible in the first line, as the 10

The therapeutic window is narrow and further clinical and/or radiological progression on the first line therapy may preclude further oncological and surgical interventions. Fit patients may benefit from a triplet of 5-FU, oxaliplatin, and irinotecan (FOLFOXIRI). However, this is a toxic regimen, and older or less fit patients are more commonly offered a doublet of 5-FU and either oxaliplatin or irinotecan. There may be an additional value when the chemotherapy is combined with antibodies targeting VEGF or, for those tumors expressing wild type KRAS, the EGF receptor.

But maybe the most valuable setting for the patient with upfront non-resectable tumor burden, would be before any treatment has started.

Up to 50% of patients with colorectal cancer will develop liver metastases either synchronous or metachronous in relation to the detection of the primary tumor[2]. The mainstay of treatment today is a combination of resection +/-ablation of metastases, with or without preoperative liver volume augmentation and chemotherapy sometimes in combination with antibodies[3].

A number of negative prognostic factors have been identified both regarding the tumor growth but also in the pattern of oncogens in the tumors[4]. Still, one of the most important factors is the response of the metastases to chemotherapy both radiologically but also in reduction of tumor markers (CEA, CA19/9)[5, 6].

Still we have very little knowledge if the metastases are going to respond to the therapy given or not. Tumor with KRAS mutation will not respond to Erbitux treatment, and mucinous tumors are usually more resistant to any chemotherapy[7].

Different models have been explored to evaluate tumor specific response to treatment, but most are slow or have shown mixed results[8]. Today, mouse patient-derived xenograft (PDX) model is the most used and validated to predict response to therapy, but evaluation of oncological therapy takes months [9]. Therefore, the mouse PDX model cannot be used for clinical decision-making. Organoid cultures using patient-derived cancers is a well-used in vitro screening tool, with promising results for different tumors[10]. Organoids maintain the genetic characteristics of the original tumor tissue. Still, these models are slow when it comes to evaluating patients' tissue for treatment decisions and lacks the ability to evaluate metastatic or angiogenic potentials.

Recently zebrafish embryos have been used as avatars for human cancer, first in hematogenous cancers but lately also in solid cancers like PDAC, breast cancer and colorectal cancer[11-14].

The model has several advantages, the strongest is response evaluation only 3-5 days after the tumor tissue is implanted in the embryos. The embryos are transparent so tumor growth and spread can be visualized in detail and quantified in a semi-automatic manner[15]. As the zebra fish embryos own immune system does not respond until day 8 days [14], why the immune response against the tumor comes from the patient's own immune cells, this is also the reason why xenograft engraftment works in this model. On the other hand. So far, biopsy tissue is not enough, but at least a cubic centimetre of tumor tissue is needed to generate these avatars. For this reason, needle biopsies are not providing enough material but resected liver tumor tissues are needed in the current protocols.

In zebrafish embryos, colorectal cancer cells have been shown to grow and response evaluation of different chemotherapy combinations have been successful with very good correlation to the response in humans[14]. Clinical studies on colorectal liver metastases have so far not been performed.

Fish are housed at an average temperature of 28 °C in a recirculating system with a 14:10 h light to dark cycle. Zebrafish fertilized eggs are obtained by natural mating of wild-type AB strain at our facilities and the developing embryos are staged in incubator at 28 °C according to Kimmel et al[19]. Before any procedure, embryos will be anesthetized in 0.02% tricaine. The tumor tissue taken from the surgical specimen by the histopathologist is cryopreserved by submerging the tissue in cryotubes containing cryopreservation medium, adding the tubes to a cryobox and placing the box in a -80 degrees freezer for at least 24 hours. The tube with tissue is then transported on dry ice to the zebrafish laboratory where the tissue will be thawed, washed and incubated in a protease mix within a mechanical disaggregation device (GentleMACS), to produce a single cell suspension from the tissue. The suspension is filtered and incubated for 30 min in 40 μg/mL CM-Dil in phosphate buffered saline (PBS), followed by centrifugation, and washing with PBS. The labeled cells are then resuspended in implantation medium and injected using thin glass capillary needles into the subcutaneous perivitelline compartment of 2-days old zebrafish embryos. Successfully implanted zebrafish embryos are then transferred to embryo medium containing the drugs under investigation (e.g. the drugs that could be considered for treatment of the patient donating the sample) and treated for three days. Images of the tumors are acquired both immediately after transplantation and following the three-day treatment period, and an additional image of the main metastatic site in the zebrafish embryo is acquired after the three-day treatment period to evaluate the metastatic capabilities of the cells. Treatment outcome will be evaluated as change in tumor volume between day 3 and day 0 in the treatment group compared to the vehicle control group (percent), and a significantly stronger reduction of tumor volumes in the treatment group will be considered as a positive treatment outcome. Evidence of a pro-metastatic phenotype will be derived from the number of cells found at the metastatic site in the zebrafish embryos three days after implantation. Cut-off levels for how many metastasized cells are required to predict likely metastatic progression in the patient will be evaluated in the first 10-20 patients included as such information is not currently available from other sources of information.

ELIGIBILITY:
Inclusion Criteria:

Confirmed or suspected diagnosis of colorectal liver metastasis Age 18 years or older ECOG 0-2 Patient can understand verbal and written information -

Exclusion Criteria:

Age less than 18 years ECOG >2 Patient is not able to understand the verbal and written information

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-05-17 (Actual); Primary Completion 2024-03-14 (Estimated); Study Completion 2025-03-14 (Estimated)

PRIMARY OUTCOMES:
Successful tumour growth in zebra fish embryos | In each embryo within 3 days
  % of implanted tumour that grow in zebrafish embryos
Response evaluation of different combinations of chemotherapy in zebra fish embryos implanted with colorectal liver metastatic tissue | In each embryo within 3 days
  The relative tumour area between the time of implantation and day 3 in each zebrafish embryo

CONTACTS AND LOCATIONS:
Overall Officials: Bärbel Jung, PhD, Study Director — University hospital Linkoing
Locations (1):
- Per Sandström, Linköping, Östergötland County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
Anonymous data will be available

REFERENCES:
- [Background] Lievre A, Bachet JB, Boige V, Cayre A, Le Corre D, Buc E, Ychou M, Bouche O, Landi B, Louvet C, Andre T, Bibeau F, Diebold MD, Rougier P, Ducreux M, Tomasic G, Emile JF, Penault-Llorca F, Laurent-Puig P. KRAS mutations as an independent prognostic factor in patients with advanced colorectal cancer treated with cetuximab. J Clin Oncol. 2008 Jan 20;26(3):374-9. doi: 10.1200/JCO.2007.12.5906. PMID 18202412
- [Background] de Jong MC, Pulitano C, Ribero D, Strub J, Mentha G, Schulick RD, Choti MA, Aldrighetti L, Capussotti L, Pawlik TM. Rates and patterns of recurrence following curative intent surgery for colorectal liver metastasis: an international multi-institutional analysis of 1669 patients. Ann Surg. 2009 Sep;250(3):440-8. doi: 10.1097/SLA.0b013e3181b4539b. PMID 19730175
- [Background] Padmanabhan C, Nussbaum DP, D'Angelica M. Surgical Management of Colorectal Cancer Liver Metastases. Surg Oncol Clin N Am. 2021 Jan;30(1):1-25. doi: 10.1016/j.soc.2020.09.002. PMID 33220799
- [Background] Kawaguchi Y, Lillemoe HA, Vauthey JN. Gene mutation and surgical technique: Suggestion or more? Surg Oncol. 2020 Jun;33:210-215. doi: 10.1016/j.suronc.2019.07.004. Epub 2019 Jul 18. PMID 31351766
- [Background] Hatano E, Okuno M, Nakamura K, Ishii T, Seo S, Taura K, Yasuchika K, Yazawa T, Zaima M, Kanazawa A, Terajima H, Kaihara S, Adachi Y, Inoue N, Furumoto K, Manaka D, Tokka A, Furuyama H, Doi K, Hirose T, Horimatsu T, Hasegawa S, Matsumoto S, Sakai Y, Uemoto S. Conversion to complete resection with mFOLFOX6 with bevacizumab or cetuximab based on K-ras status for unresectable colorectal liver metastasis (BECK study). J Hepatobiliary Pancreat Sci. 2015 Aug;22(8):634-45. doi: 10.1002/jhbp.254. Epub 2015 Apr 29. PMID 25926024
- [Background] Rehman AH, Jones RP, Poston G. Prognostic and predictive markers in liver limited stage IV colorectal cancer. Eur J Surg Oncol. 2019 Dec;45(12):2251-2256. doi: 10.1016/j.ejso.2019.06.038. Epub 2019 Jun 27. PMID 31279594
- [Background] Reynolds IS, Cromwell PM, Hoti E. Clinicopathological characteristics and survival outcomes for patients with mucinous colorectal cancer liver metastases undergoing hepatic resection: A systematic review and meta-analysis. Am J Surg. 2021 Sep;222(3):529-535. doi: 10.1016/j.amjsurg.2021.02.031. Epub 2021 Mar 3. PMID 33750573
- [Background] Mauri G, Durinikova E, Amatu A, Tosi F, Cassingena A, Rizzetto F, Buzo K, Arcella P, Aquilano MC, Bonoldi E, Marsoni S, Siena S, Bardelli A, Sartore-Bianchi A, Arena S. Empowering Clinical Decision Making in Oligometastatic Colorectal Cancer: The Potential Role of Drug Screening of Patient-Derived Organoids. JCO Precis Oncol. 2021 Jul 21;5:PO.21.00143. doi: 10.1200/PO.21.00143. eCollection 2021 Jul. No abstract available. PMID 34327296
- [Background] Costa B, Estrada MF, Mendes RV, Fior R. Zebrafish Avatars towards Personalized Medicine-A Comparative Review between Avatar Models. Cells. 2020 Jan 25;9(2):293. doi: 10.3390/cells9020293. PMID 31991800
- [Background] Yang H, Sun L, Liu M, Mao Y. Patient-derived organoids: a promising model for personalized cancer treatment. Gastroenterol Rep (Oxf). 2018 Nov;6(4):243-245. doi: 10.1093/gastro/goy040. Epub 2018 Oct 9. No abstract available. PMID 30430011
- [Background] Yao Y, Wang L, Wang X. Modeling of Solid-Tumor Microenvironment in Zebrafish (Danio Rerio) Larvae. Adv Exp Med Biol. 2020;1219:413-428. doi: 10.1007/978-3-030-34025-4_22. PMID 32130712
- [Background] Mercatali L, La Manna F, Groenewoud A, Casadei R, Recine F, Miserocchi G, Pieri F, Liverani C, Bongiovanni A, Spadazzi C, de Vita A, van der Pluijm G, Giorgini A, Biagini R, Amadori D, Ibrahim T, Snaar-Jagalska E. Development of a Patient-Derived Xenograft (PDX) of Breast Cancer Bone Metastasis in a Zebrafish Model. Int J Mol Sci. 2016 Aug 22;17(8):1375. doi: 10.3390/ijms17081375. PMID 27556456
- [Background] Di Franco G, Usai A, Funel N, Palmeri M, Montesanti IER, Bianchini M, Gianardi D, Furbetta N, Guadagni S, Vasile E, Falcone A, Pollina LE, Raffa V, Morelli L. Use of zebrafish embryos as avatar of patients with pancreatic cancer: A new xenotransplantation model towards personalized medicine. World J Gastroenterol. 2020 Jun 7;26(21):2792-2809. doi: 10.3748/wjg.v26.i21.2792. PMID 32550755
- [Background] Fior R, Povoa V, Mendes RV, Carvalho T, Gomes A, Figueiredo N, Ferreira MG. Single-cell functional and chemosensitive profiling of combinatorial colorectal therapy in zebrafish xenografts. Proc Natl Acad Sci U S A. 2017 Sep 26;114(39):E8234-E8243. doi: 10.1073/pnas.1618389114. Epub 2017 Aug 23. PMID 28835536
- [Background] Lubin A, Otterstrom J, Hoade Y, Bjedov I, Stead E, Whelan M, Gestri G, Paran Y, Payne E. A versatile, automated and high-throughput drug screening platform for zebrafish embryos. Biol Open. 2021 Sep 15;10(9):bio058513. doi: 10.1242/bio.058513. Epub 2021 Sep 2. PMID 34472582